CLINICAL TRIAL: NCT05128890
Title: Evaluation of Resection Techniques for Pancreatic Tumors
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 028.HPB.2016.D
Record Dates: First submitted 2019-08-12; First posted 2021-11-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Surgery; Liver Tumor; Pancreas Tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Pancreatic Neoplasms | interventions — Pancreatic Hormones

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Resection techniques for pancreatic and liver tumors — to compare open versus minimally invasive pancreatic resection techniques and analyze the different outcome variables from the clinical standpoint
  Other Names: minimally invasive pancreatic resection techniques

SUMMARY:
The objective of this study is to compare open and minimally invasive pancreatic and liver resection techniques and analyze the different outcome variables from the clinical standpoint.

The plan is to investigate patient survival, length of stay, complication rates, operative time, transfusion rate, 30 and 90-day readmission rate, and hospital charges.

DETAILED DESCRIPTION:
The plan is to conduct a retrospective chart review of patients who have undergone pancreatic and liver resection by using Meditech and Epic. A non-identified database will be created after retrospectively reviewing each patient case involving pancreatic or liver resection at MDMC. The study period will start in January 2006 until December 2020. Variables will include demographics, clinical disease diagnoses, and operative parameters as well as indirect charges from the hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have undergone pancreatic or liver resection surgeries from January 2006 until December 2020 at Methodist Dallas Medical Center (MDMC)
* Patients 18 years old or older

Exclusion Criteria:

* Patients that have not undergone pancreatic resection surgeries
* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pancreatic or liver resection surgeries from January 2006 until December 2020 at Methodist Dallas Medical Center (MDMC)
Sampling Method: Non-Probability Sample
Enrollment: 431 (Estimated)
Dates: Start 2016-04-16 (Actual); Primary Completion 2026-04-26 (Estimated); Study Completion 2026-04-26 (Estimated)

PRIMARY OUTCOMES:
Patient Survival | through study completion, an average of 1 year
  It will be calculated in days.Minimally invasive techniques are being adopted for complex pancreatic and liver surgery and there is a need to understand if these techniques are advantageous to the patient, if the cost is justified and if the risks are acceptable when compared to the gold standard open surgery.
Length of stay | Up to 1 year
  It will be calculated in days. The days stayed in hospital post-procedure.
Complication rates | through study completion, an average of 1 year
  Patient may visit physician or hospital for any symptoms or may need hospitalizations.
Operative time | up to 10 hours
  The time required for the procedure.
Transfusion rate | through study completion, an average of 1 year
  If any post-procedure transfusion required, will be recorded.
30 and 90 day readmission rate | through study completion, an average of 1 year
  After the procedure any hospital admissions up to 30 days will be recorded.
Hospital charges | through study completion, an average of 1 year
  The hospital charges for the procedure will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Mejia, M.D., Principal Investigator — The Liver Institute, Methodist Dallas Medical Center
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No